CLINICAL TRIAL: NCT01434342
Title: Feasibility of Delivering a Quitline Based Smoking Cessation Intervention in Lung Cancer Patients Receiving Outpatient Treatment: A Pilot Study
Brief Title: Feasibility of Delivering a Quitline Based Smoking Cessation Intervention in Cancer Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB000019384; U10CA081851 (NIH); REBACCCWFU 99211 (Other: NCI)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer; Tobacco Use Disorder; Breast Cancer; Colorectal Cancer; Prostate Cancer
Keywords: stage IA non-small cell lung cancer; stage IB non-small cell lung cancer; stage IIA non-small cell lung cancer; stage IIB non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; limited stage small cell lung cancer; tobacco use disorder; Breast Cancer; Cervical Cancer; head & neck cancer; Prostate Cancer; All histologies
MeSH Terms: conditions — Lung Neoplasms; Tobacco Use Disorder; Breast Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Uterine Cervical Neoplasms; Head and Neck Neoplasms | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I - Quitline (Experimental): Participants receive a letter from their physician advising them to quit smoking, and undergo a 15-30-minute smoking-cessation counseling session by a trained research staff.
  The participants are educated and motivated about the importance of quitting smoking, and cancer-specific quitting issues. They will be called by Quitline in 2-3 days and receive a fact sheet about benefits of SC for cancer patients.
  Participants receive 8 weeks of nicotine replacement patches and up to 5 proactive telephone calls over a 12-week period.
  Participants also learn behavioral tips and coping skills.
  Interventions: Drug: Nicotine Replacement Patch
- Arm II - Usual Care (No Intervention): Participants receive a letter from their physician advising them to quit smoking, the importance of quitting smoking for cancer patients, and a copy of the National Cancer Institute's "Clearing the Air" smoking cessation booklet. Participants also receive standard of care from their oncology and other treatment providers which may or may not include nicotine replacement therapy.

INTERVENTIONS:
Drug: Nicotine Replacement Patch — Study participants will receive a baseline assessment after they consent to participate and before randomization. The intervention period will last 12 weeks (approximately 1 week for the in-office intervention and 12 weeks for all components of the Quitline intervention- telephone counseling and habitrol patches). Follow-up assessments will be administered at 3, 6, 12, & 24 weeks after the date of the in-person intervention (for Quitline Intervention group) or the provision of the physician letter (for the Usual Care Plus group).
  Other Names: Nicotine patch; Habitrol patch
  Arms: Arm I - Quitline

SUMMARY:
RATIONALE: Continued smoking after a cancer diagnosis has important health consequences beyond the risks associated with smoking in the general population. Smoking reduces the efficacy of cancer treatments including surgery, radiation and chemotherapy. Despite the negative consequences, it is estimated that between 15-75% of patients with cancer continue to smoke after their cancer diagnosis. Lung, breast, prostate, colorectal, bladder, head & neck, and cervical cancer patients were chosen because there is evidence of potential clinical benefit associated with quitting smoking in all of these populations and they represent a mix of both smoking and non-smoking related cancers.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the feasibility of delivering a Quitline based smoking cessation intervention to cancer patients in an outpatient setting. To achieve this, we will deliver the intervention to cancer patients in the surgery, radiation and medical oncology departments of participating Community Clinical Oncology Program (CCOP) sites. Following the intervention, we will assess participant, CRA (Clinical Research Associate) Counselor and Quitline staff ratings of acceptability, resources required to deliver the intervention, protocol fidelity, and participant recruitment, retention and adherence.

Secondary

* To obtain a preliminary estimate of the quit rate (as defined by 7-day point-prevalence abstinence) in intervention and control groups. To accomplish this aim, following the intervention we will collect confirmed smoking status data for intervention and control subjects. We will also obtain a preliminary estimate of the treatment effect (difference in quit rates between the two groups) and the standard deviation to better determine the sample size for a future trial.
* To evaluate primary patient reported outcomes, including quality of life (quantified by the FACT-G and for lung cancer patients only the FACT-L other concerns questions and the EORTC QLQ LC13), perceived life stress (quantified by the Perceived Stress Scale), and depression (quantified by the CESD-10), in cancer patients in the intervention and control groups.
* To refine the recruitment and intervention protocols using data collected from participants, Clinical Research Associate (CRA) Counselor, and Quitline staff to increase acceptability and improve retention in future trials.

OUTLINE: This is a multicenter study. Participants are stratified according to time since diagnosis (< 3 months vs ≥ 3 months), treatment status (ongoing vs completed), and cigarette smoking (≤ 10 per day vs ≥ 11 per day). Patients are randomized to 1 of 2 intervention arms.

* Arm I (intervention): Participants receive a letter from their physician advising them to quit smoking, and undergo a 15-30-minute smoking-cessation counseling session by a trained research staff. During the counseling session, participants are educated and motivated about the importance of quitting smoking, and cancer-specific quitting issues such as managing the stressors associated with cancer diagnosis and treatment. They are also told to expect a call from the Quitline in 2-3 days and receive a fact sheet about benefits of smoking cessation for cancer patients. Participants receive 8 weeks of nicotine replacement patches and up to 5 proactive telephone calls over a 12-week period. Calls are scheduled at convenient times for the participants and at relapse-sensitive intervals including; an initial planning and assessment call, a quit date call, a follow-up call 7 days after the participant's quit date, and 2 additional calls at 2-3-week intervals. Participants are also encouraged to utilize the Quit for Life Web Coach, an interactive web program application that guides them to build online quit plans, set quit dates, and track their progress toward quitting. Participants also learn behavioral tips and coping skills by interacting with others in topic-based discussion forums and community support programs.
* Arm II (standard of care): Participants receive a letter from their physician advising them to quit smoking, the importance of quitting smoking for cancer patients, and a copy of the National Cancer Institute's "Clearing the Air" smoking cessation booklet. Participants also receive standard of care from their oncology and other treatment providers which may or may not include nicotine replacement therapy.

Participants on the intervention arm complete the Smoking Assessment, Smoking Cessation Self-Efficacy, the Brief Smoking Consequences, the Functional Assessment of Cancer Therapy-Lung Cancer (FACT-L), the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire LC-13, the Perceived Stress Scale, the Center for Epidemiologic Studies Short Depression Scale (CESD-10 Depression), and the Follow up Smoking Assessment questionnaires at baseline and at 6, 12, and 24 weeks.

Participants, on the intervention arm, undergo saliva sample collection at baseline and at 12 and 24 weeks for cotinine level analysis.

ELIGIBILITY:
Inclusion Criteria:

1. AJCC Stages 0, I, II, & III lung, breast, prostate, colorectal, bladder, head & neck, and cervical cancers (all histologies).
2. Reports smoking any amount in the last 7 days.
3. Scheduled to receive or currently receiving surgery, radiation or chemotherapy OR have received one or more of the following in the last 6 months surgery, last radiation treatment or last chemotherapy treatment.
4. 18 years of age or older
5. KPS of 70-100
6. Ability to understand and the willingness to sign a written informed consent document.
7. Willing to consider quitting smoking

Exclusion Criteria:

1. Unstable cardiac disease - defined as congestive heart failure, unstable angina, serious arrhythmias, or Myocardial Infarction in the past month.
2. Current use or planned use of varenicline (Chantix), Zyban, Buproprion or any other nicotinic receptor agonist (Patients that discontinue use of these type drugs within 7 days are eligible.)
3. Current probable alcohol abuse as defined by more than 5 drinks per day for men and 4 drinks per day for women and a Alcohol Use Disorders Identification Test (AUDIT) score > 8.

   If patient answers "no" to 5 drinks per day for men and 4 drinks per day for women the patient is eligible. AUDIT assessment does not need to be administered.

   If patient answers "yes " to 5 drinks per day for men and 4 drinks per day for women the AUDIT assessment must be administered. If AUDIT score is > 8 patient is not eligible.
4. Use of illegal drugs or use of prescription medications for non-medical reasons in the past month.
5. Current use of chewing, dipping and pipe tobacco, or cigars.
6. Patient does not have regular access to a telephone to receive Quitline calls lasting 15-30 minutes.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to nicotine replacement therapy.
8. Active Peptic Ulcer Disease
9. Uncontrolled intercurrent illness including, but not limited to, ongoing, psychiatric illness/social situations that would limit compliance with study requirements.
10. Due to unknown risks and potential harm to the unborn fetus, sexually active women of childbearing potential must use a reliable method of birth control while participating in this study. Reliable methods of birth control are: abstinence (not having sex), oral contraceptives, intrauterine device (IUD), DepoProvera, tubal ligation, or vasectomy of the partner (with confirmed negative sperm counts) in a monogamous relationship (same partner). An acceptable, although less reliable, method involves the careful use of condoms and spermicidal foam or gel and/or a cervical cap or sponge. We encourage you to discuss this issue further with your doctors if you have any questions.
11. If you are pregnant, should become pregnant or suspect you are pregnant prior to or while participating in this study, you should inform your study physician immediately. Nicotine replacement therapy has the potential for teratogenic or abortifacient effects and is classified as a FDA Pregnancy category D drug. The U.S. Clinical Practice Guideline states that pregnant smokers should be encouraged to quit without medication based on insufficient evidence of effectiveness and hypothetical concerns with safety. Pregnant women enrolled in the study and randomized to the Quitline group intervention should participate in the Quitline intervention but not receive the nicotine replacement therapy.
12. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nicotine replacement therapy, breastfeeding women are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2014-06-01 (Actual); Study Completion 2015-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Weaver, PhD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- W F Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Quitline Based Smoking Cessation — https://www.clinicaltrials.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants are recruited from NCI CCOP sites
Groups:
- Quitline: Participants receive a letter from their physician advising them to quit smoking, and undergo a 15-30-minute smoking-cessation counseling session by a trained research staff. The participants are educated and motivated about the importance of quitting smoking, and cancer-specific quitting issues. They will be called by Quitline in 2-3 days and receive a fact sheet about benefits of SC for cancer patients. Participants receive 8 weeks of nicotine replacement patches and up to 5 proactive telephone calls over a 12-week period. Participants also learn behavioral tips and coping skills.
  Nicotine Replacement Patch: Study participants will receive a baseline assessment after they consent to participate and before randomization. The intervention period will last 12 weeks (approximately 1 week for the in-office intervention and 12 weeks for all components of the Quitline intervention- telephone counseling and habitrol patches). Follow-up assessments will be administered at 3, 6, 12, & 24 we
- Usual Care: Participants receive a letter from their physician advising them to quit smoking, the importance of quitting smoking for cancer patients, and a copy of the National Cancer Institute's "Clearing the Air" smoking cessation booklet. Participants also receive standard of care from their oncology and other treatment providers which may or may not include nicotine replacement therapy.
Period: Overall Study
Arm/Group | Quitline | Usual Care
Started | 98 | 48
Completed | 50 | 31
Not Completed | 48 | 17

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Arm I - Quitline: Participants receive a letter from their physician advising them to quit smoking, and undergo a 15-30-minute smoking-cessation counseling session by a trained research staff. The participants are educated and motivated about the importance of quitting smoking, and cancer-specific quitting issues. They will be called by Quitline in 2-3 days and receive a fact sheet about benefits of SC for cancer patients. Participants receive 8 weeks of nicotine replacement patches and up to 5 proactive telephone calls over a 12-week period. Participants also learn behavioral tips and coping skills.
  Nicotine Replacement Patch: Study participants will receive a baseline assessment after they consent to participate and before randomization. The intervention period will last 12 weeks (approximately 1 week for the in-office intervention and 12 weeks for all components of the Quitline intervention- telephone counseling and habitrol patches). Follow-up assessments will be administered at 3, 6, 12, & 24 we
- Arm II: Participants receive a letter from their physician advising them to quit smoking, the importance of quitting smoking for cancer patients, and a copy of the National Cancer Institute's "Clearing the Air" smoking cessation booklet. Participants also receive standard of care from their oncology and other treatment providers which may or may not include nicotine replacement therapy.
- Total: Total of all reporting groups
Arm/Group | Arm I - Quitline | Arm II | Total
Number analyzed (Participants) | 98 | 48 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 69 | 35 | 104
  >=65 years | 29 | 13 | 42
Age, Continuous [Median (Full Range); unit: years] | 57 [22 to 75] | 58 [26 to 86] | 57 [22 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 36 | 109
  Male | 25 | 12 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 96 | 48 | 144
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 8 | 27
  White | 77 | 40 | 117
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 98 | 48 | 146

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of a Smoking Cessation Intervention Among Cancer Patients
Description: The primary feasibility measures are retention and adherence. This outcome, retention, is the percentage of patient who remain in the study for 24 weeks.
Time Frame: 24 Weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I - Quitline | Arm II - Usual Care
Number analyzed (Participants) | 98 | 48
Participants | 55 | 33

2. Primary Outcome: Adherence
Description: Adherence is measured by the percentage of randomized participants who have a Quitline call. Note that this outcome is only defined for the Intervention arm
Time Frame: 24 weeks
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I - Quitline | Arm II - Usual Care
Number analyzed (Participants) | 98 | 0
Participants | 81 |

ADVERSE EVENTS:
Time Frame: 24 weeks
Description: Sample size is the number of participants with follow-up toxicity data
Arm/Group | Arm I - Quitline | Arm II - Usual Care
Serious Adverse Events (participants affected / at risk) | 14/75 | 5/37
Other Adverse Events (participants affected / at risk) | 61/75 | 33/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Quitline (N=75) | Arm II - Usual Care (N=37)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Bladder Infection (Infections and infestations) | 1 (1) | 0 (0)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal Infection (Infections and infestations) | 1 (1) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Neutrophil Count (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Thromboembolic event (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - Quitline (N=75) | Arm II - Usual Care (N=37)
Anorexia (Psychiatric disorders) | 3 (5) | 2 (3)
Anxiety (Psychiatric disorders) | 35 (74) | 15 (27)
Chest pain cardiac (Cardiac disorders) | 6 (9) | 3 (4)
Constipation (Gastrointestinal disorders) | 21 (41) | 9 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (15) | 5 (9)
Depression (Psychiatric disorders) | 26 (56) | 14 (27)
Diarrhea (Gastrointestinal disorders) | 9 (18) | 3 (3)
Dry Mouth (Skin and subcutaneous tissue disorders) | 21 (34) | 9 (17)
Dyspepsia (Gastrointestinal disorders) | 15 (30) | 7 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 39 (93) | 15 (27)
Fatigue (Metabolism and nutrition disorders) | 18 (30) | 7 (14)
Headache (Nervous system disorders) | 25 (41) | 6 (8)
Insomnia (General disorders) | 28 (58) | 11 (19)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 4 (8) | 0 (0)
Myalagia (Musculoskeletal and connective tissue disorders) | 22 (48) | 13 (28)
Nausea (Gastrointestinal disorders) | 23 (41) | 3 (5)
Nervous system disorder (Nervous system disorders) | 1 (2) | 2 (2)
Pain (General disorders) | 12 (16) | 4 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4) | 3 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 17 (17) | 4 (4)
Psychiatric disorder (Psychiatric disorders) | 4 (9) | 3 (5)
Rash masculo-papular (Skin and subcutaneous tissue disorders) | 7 (8) | 2 (2)
Skin and subcutaneous tissue (Skin and subcutaneous tissue disorders) | 8 (8) | 2 (3)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes